CLINICAL TRIAL: NCT04538989
Title: An Open-Label Multiple-Dose Study of RZ358 in Patients With Congenital Hyperinsulinism
Brief Title: An Open-Label Multiple Dose Study of RZ358 in Patients With Congenital Hyperinsulinism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rezolute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RZ358-606
Record Dates: First submitted 2020-08-21; First posted 2020-09-04 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Congenital Hyperinsulinism
Keywords: Hypoglycemia; Congenital Hyperinsulinism; Glucose Metabolism Disorders; Metabolic Diseases; Pancreatic Diseases; Digestive System Diseases; Hyperinsulinism
MeSH Terms: conditions — Congenital Hyperinsulinism; Hypoglycemia; Glucose Metabolism Disorders; Metabolic Diseases; Pancreatic Diseases; Digestive System Diseases; Hyperinsulinism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- RZ358 Cohort 1 (Experimental)
  Interventions: Drug: RZ358 Sequential Group Cohort 1
- RZ358 Cohort 2 (Experimental)
  Interventions: Drug: RZ358 Sequential Group Cohort 2
- RZ358 Cohort 3 (Experimental)
  Interventions: Drug: RZ358 Sequential Group Cohort 3
- RZ358 Cohort 4 (Experimental)
  Interventions: Drug: RZ358 Sequential Group Cohort 4

INTERVENTIONS:
Drug: RZ358 Sequential Group Cohort 1 — IV infusion for 8 weeks (3 mg/kg bi-weekly for 8 weeks)
  Arms: RZ358 Cohort 1
Drug: RZ358 Sequential Group Cohort 2 — IV infusion for 8 weeks (6 mg/kg bi-weekly for 8 weeks)
  Arms: RZ358 Cohort 2
Drug: RZ358 Sequential Group Cohort 3 — IV infusion for 8 weeks (9 mg/kg bi-weekly for 8 weeks)
  Arms: RZ358 Cohort 3
Drug: RZ358 Sequential Group Cohort 4 — IV infusion for 8 weeks (bi-weekly fixed dose-titration from 3 to 9 mg/kg for the first 4 weeks, followed by a fixed 9 mg/kg dose amount thereafter for the remaining 4 weeks)
  Arms: RZ358 Cohort 4

SUMMARY:
The objective of this trial is to evaluate the safety, tolerability and glucose-raising effects of RZ358 in patients with Congenital Hyperinsulinism (HI).

DETAILED DESCRIPTION:
There is a significant unmet medical need to develop new therapies aimed at preventing chronic recurrent hypoglycemia in congenital HI, the most common cause of persistent hypoglycemia in children. RZ358 is a human mAb that allosterically attenuates excessive insulin action on target cells. Therefore, RZ358 is ideally suited as a potential therapy for hyperinsulinism, and it is being developed to treat the hypoglycemia associated with diseases such as congenital HI. This is a Phase 2, multicenter, open label clinical study designed to assess the safety and efficacy of four progressively higher doses of RZ358 in separate groups of patients with hyperinsulinemic hypoglycemia due to Congenital HI, not adequately controlled with or without current standard of care. A screening period of up to 5 weeks will evaluate eligibility. Once enrolled, RZ358 will be administered bi-weekly over 8 weeks, and then patients will complete a post-treatment follow-up period of 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 2-45 years old (except age 12-45 in US) with an established clinical diagnosis of congenital hyperinsulinism
* Able to provide written informed consent or, as applicable, assent
* Confirmed hypoglycemia as assessed by CGM, SMBG, and clinical evaluation, during Screening
* Willingness to use contraception if of child-bearing potential

Exclusion Criteria:

* Out of range blood work for study entry
* Body Mass index outside of study entry criteria
* History of malignancy
* Clinically significant diseases, seropositivity for HIV, hepatitis B or C antibody
* Use of systemic corticosteroids within 30 days before Screening
* Known or suspected allergy to the study drug
* Recent use of an investigational drug or treatment, or participation in an investigational study
* Pregnant or lactating women
* History of drug abuse or excessive alcohol use

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-08-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (2):
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center, Fort Worth, Texas
- Bulgaria (2):
  - SHAT Children diseases "Prof. Dr. Ivan Mitov", Sofia
  - Medical University of Varna UMHAT "St. Marina", Varna
- Research Institute of the McGill University Health Centre, Monteral, Qubec, Canada
- Odense University Hospital, Odense, Denmark
- LTD "Pediatric Surgery Centre", Tbilisi, Georgia
- Magdeburg University Clinic Center (Otto-von-Guericke Universität), Magdeburg, Germany
- Israel (2):
  - Edmond & Lilly Safra's Children Hospital, Ramat Gan, Tel-Hashomer
  - Hadassah Har Hazofim MC - Division of Pediatric Endocrinology, Jerusalem
- Endocrinology research center, Moscow, Russia
- Hospital Universitari Vall d' Hebron, Barcelona, Spain
- Turkey (Türkiye) (4):
  - Adana Cukurova University Balcalı Hospital, Sarıçam, Adana
  - Hacettepe University, Çankaya, Ankara
  - SBÜ Gazi Yaşargil Eğitim ve Araştirma Hastanesi, Kayapınar, Diyarbakır
  - Erzurum City Hospital, Yakutiye, Erzurum
- Great Ormond Street Hospital, London, United Kingdom

REFERENCES:
- [Derived] Demirbilek H, Melikyan M, Iotova V, Galcheva S, Ozbek MN, Dastamani A, Kheladze N, Mazor-Aronovitch K, Clemente M, Empting S, Mohnike K, Christesen HT, Thornton PS, De Leon DD, Hood D, O'Boyle E, Roberts BK. Global, multi-center, repeat-dose, phase 2 study of RZ358 (ersodetug), an insulin receptor antibody, for congenital hyperinsulinism. Med. 2025 Jun 13;6(6):100611. doi: 10.1016/j.medj.2025.100611. Epub 2025 Mar 18. PMID 40107271

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sites were recruited based on cHI professional expertise and sufficient patient panels and advocacy referrals.
Pre-assignment Details: NA; open-label study
Period: Overall Study
Arm/Group | RZ358 Cohort 1 | RZ358 Cohort 2 | RZ358 Cohort 3 | RZ358 Cohort 4
Started | 4 | 8 | 8 | 3
Completed | 4 | 8 | 8 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RZ358 Cohort 1 | RZ358 Cohort 2 | RZ358 Cohort 3 | RZ358 Cohort 4 | Total
Number analyzed (Participants) | 4 | 8 | 8 | 3 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 7 | 8 | 3 | 22
  Between 18 and 65 years | 0 | 1 | 0 | 0 | 1
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.8 (4.35) | 9.3 (6.88) | 5.8 (5.12) | 4.0 (2.00) | 6.7 (5.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 3 | 1 | 13
  Male | 0 | 3 | 5 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 6 | 8 | 3 | 21
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 4 | 6 | 7 | 3 | 20
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Turkey | 0 | 3 | 4 | 0 | 7
  United States | 0 | 1 | 0 | 0 | 1
  Denmark | 0 | 1 | 0 | 0 | 1
  United Kingdom | 0 | 1 | 1 | 0 | 2
  Georgia | 1 | 0 | 0 | 0 | 1
  Israel | 0 | 1 | 0 | 0 | 1
  Bulgaria | 3 | 0 | 0 | 0 | 3
  Germany | 0 | 0 | 1 | 0 | 1
  Russia | 0 | 0 | 2 | 3 | 5
  Spain | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Median of Average Daily Percent Time Within a Glucose Target Range of 70-180 mg/dL (3.9-10 mmol/L) by CGM at Baseline (BL) and End of Treatment (EOT)
Description: The median of average daily percent time within the glucose target range 70-180 mg/dL (3.9-10 mmol/L) by CGM at Baseline and End of Treatment (EOT) is reported.
Time Frame: 8 weeks
Population: Per Protocol Population
Measure: Median (95% Confidence Interval); unit: Daily Percent Time
Groups:
- RZ358 Pooled: RZ358 Total Participants
Arm/Group | RZ358 Cohort 1 | RZ358 Cohort 2 | RZ358 Cohort 3 | RZ358 Cohort 4 | RZ358 Pooled
Number analyzed (Participants) | 4 | 8 | 7 | 3 | 22
Daily Percent Time
  Median of Average Daily Percent Time in 70-180 mg/dL at BL | 81.7 [70.5 to 92.5] | 72.9 [67.5 to 80.9] | 83.4 [43.2 to 94.8] | 59.3 [25.7 to 110] | 76.9 [65.3 to 80.7]
  Median of Average Daily Percent Time in 70-180 mg/dL at 8 weeks (EOT) | 84.8 [71.6 to 100.3] | 78.5 [61.1 to 88.6] | 82.9 [67.1 to 91.6] | 70.8 [50.9 to 93.9] | 79.1 [72.0 to 83.9]

2. Primary Outcome: Median Percent Change of Average Daily Percent Time Within a Glucose Target Range of 70-180 mg/dL (3.9-10 mmol/L) by CGM From Baseline (BL)
Description: The average daily percent time within the glucose target range (70-180 mg/dL) is compared from baseline to end of treatment (EOT) and the median percent change of that difference is reported.
Time Frame: 8 weeks
Population: Per Protocol Population
Measure: Median (95% Confidence Interval); unit: Percent Change
Arm/Group | RZ358 Cohort 1 | RZ358 Cohort 2 | RZ358 Cohort 3 | RZ358 Cohort 4 | RZ358 Pooled
Number analyzed (Participants) | 4 | 8 | 7 | 3 | 22
Percent Change | 6.19 [-2.80 to 13.6] | 0.31 [-19.7 to 24.2] | 5.52 [-82.3 to 215.2] | 9.07 [-29.6 to 48.4] | 4.59 [-16.7 to 65.1]

3. Primary Outcome: Repeat Dose Pharmacokinetics of RZ358
Description: All patients who received RZ358 and for whom the primary PK data was considered to be sufficient and interpretable were to be included in the PK analyses. Individual and mean plasma concentration data is summarized descriptively at the specified timepoints. The results of this study may be combined with those of other studies for analysis and modeling (e.g., population PK and PK-PD), and therefore the PK parameters are reported separately, as part of an iterative population PK approach.
Time Frame: Pre dose Weeks 1,3,5,7, 1-hr post dose Week 1 and Week 7, and Follow up on Days 14, Day 28, Day 42, and Day 105
Population: PK Population; Data from Cohort 1, 2 and 4 was not collected during Pre-dose Week 1.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | RZ358 Cohort 1 | RZ358 Cohort 2 | RZ358 Cohort 3 | RZ358 Cohort 4 | RZ358 Pooled
Number analyzed (Participants) | 4 | 8 | 8 | 3 | 23
ng/mL
  Pre dose Week 1: number analyzed (Participants) | 0 | 0 | 8 | 0 | 8
  Pre dose Week 1 |  |  | 55648 [55648 to 55648] |  | 55648 [55648 to 55648]
  Post dose (1hr) Wk1/D1 | 29093 [1308 to 96685] | 120368 [74257 to 190700] | 164047 [73398 to 250230] | 43593 [36330 to 53742] | 89333 [1308 to 250230]
  Pre dose Week 3 | 38951 [15363 to 83824] | 28397 [21187 to 35857] | 41512 [19816 to 60351] | 8961 [7244 to 10613] | 28999 [7244 to 83824]
  Pre dose Week 5 | 20692 [20692 to 20692] | 82646 [36116 to 376850] | 74457 [51606 to 99696] | 34243 [26150 to 42212] | 64808 [20692 to 376850]
  Pre dose Week 7 | 31902 [31902 to 31902] | 56919 [29669 to 82349] | 95721 [55202 to 123120] | 55532 [48740 to 68459] | 67823 [29669 to 123120]
  Post dose (1hr) Week 7 | 94593 [94593 to 94593] | 178090 [123230 to 245640] | 280843 [141480 to 527410] | 245905 [181540 to 434760] | 217295 [94593 to 527410]
  Follow-Up Day 14/EOT | 59542 [42139 to 76282] | 70990 [48766 to 99871] | 105005 [78798 to 129580] | 110134 [93403 to 127370] | 82683 [42139 to 129580]
  Follow-up Day 28 | 46751 [27504 to 125040] | 39385 [26997 to 59121] | 63201 [45579 to 108180] | 52039 [48235 to 57834] | 50125 [26997 to 125040]
  Follow-up Day 42 | 23166 [14390 to 29879] | 24226 [13552 to 37256] | 43034 [26741 to 60868] | 37394 [30944 to 50353] | 31066 [13552 to 60868]
  Follow-up Day 105 | 2307 [1201 to 3412] | 4231 [1105 to 15651] | 9269 [3743 to 14616] | 4194 [3297 to 6469] | 4857 [1105 to 15651]

4. Secondary Outcome: Median of Average Weekly Overall, Moderate, and Severe Hypoglycemia Events by SMBG at Baseline (BL) and End of Treatment (EOT)
Description: The median of average weekly number of overall hypoglycemia events (<70 mg/dL [3.9mmol/L], moderate hypoglycemia events (<60 mg/dL [3.3 mmol/L] and severe hypoglycemia events (<50 mg/dL [2.8mmol/L]) by SMBG at baseline (BL) and end of treatment (EOT) is reported.
Time Frame: 8 weeks
Population: Per Protocol Population; For efficacy outcomes, the PP Population included 20 participants for BGM-based glycemic endpoints due to endpoint-specific exclusions. One participant in Cohort 1 and one in Cohort 4 were excluded from the PP population BGM-based analyses because they failed to meet pre-specified minimum testing frequency by glucometer. One participant in Cohort 3 was also excluded from the PP population BGM analyses for stopping background SOC therapy after starting RZ358 in the study
Measure: Median (95% Confidence Interval); unit: Hypoglycemia Events
Arm/Group | RZ358 Cohort 1 | RZ358 Cohort 2 | RZ358 Cohort 3 | RZ358 Cohort 4 | RZ358 Pooled
Number analyzed (Participants) | 3 | 8 | 7 | 2 | 20
Hypoglycemia Events
  Median Overall Hypoglycemia Events (<70 mg/dL; <3.9 mmol/L) at BL | 10.1 [2.46 to 17.7] | 12.5 [2.94 to 28.9] | 13.0 [9.15 to 23.2] | 9.30 [-6.02 to 24.6] | 11.5 [9.43 to 19.5]
  Median Overall Hypoglycemia Events (<70 mg/dL; <3.9 mmol/L) at 8 Weeks (EOT) | 9.92 [1.85 to 15.4] | 6.60 [2.40 to 15.6] | 1.87 [-2.70 to 12.8] | 7.60 [-19.0 to 34.2] | 5.00 [4.12 to 10.7]
  Median Moderate Hypoglycemia Events (<60 mg/dL; <3.3 mmol/L) at BL | 3.06 [-0.84 to 8.05] | 6.69 [0.158 to 21.2] | 9.00 [4.18 to 19.0] | 3.69 [-5.08 to 12.5] | 5.99 [4.80 to 13.7]
  Median Moderate Hypoglycemia Events (<60 mg/dL; <3.3 mmol/L) at 8 Weeks (EOT) | 6.42 [-1.52 to 12.9] | 3.17 [0.945 to 9.00] | 0.47 [-3.13 to 10.1] | 4.18 [-4.40 to 12.8] | 2.75 [2.08 to 6.89]
  Median Severe Hypoglycemia Events (<50 mg/dL; <2.8 mmol/L) at BL | 1.31 [0.32 to 2.58] | 2.59 [-0.71 to 10.4] | 3.50 [-0.20 to 8.66] | 0.91 [-4.24 to 6.05] | 1.90 [1.35 to 6.10]
  Median Severe Hypoglycemia Events (<50 mg/dL; <2.8 mmol/L) at 8 Weeks (EOT) | 1.17 [-3.47 to 6.97] | 0.94 [0.15 to 2.34] | 0.00 [-0.74 to 2.77] | 0.52 [0.27 to 0.77] | 0.49 [0.45 to 1.88]

5. Secondary Outcome: Median Percent Change of Average Weekly Overall, Moderate, and Severe Hypoglycemia Events by SMBG From Baseline (BL)
Description: The average weekly number overall hypoglycemia events (<70 mg/dL [3.9mmol/L], moderate hypoglycemia events (<60 mg/dL [3.3 mmol/L] and severe hypoglycemia events (<50 mg/dL [2.8mmol/L]) by SMBG is compared from baseline (BL) to end of treatment (EOT) and the median percent changes of those differences are reported.
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Percent Change
Arm/Group | RZ358 Cohort 1 | RZ358 Cohort 2 | RZ358 Cohort 3 | RZ358 Cohort 4 | RZ358 Pooled
Number analyzed (Participants) | 3 | 8 | 7 | 2 | 20
Percent Change
  Median Percent Change of Overall Hypoglycemia Events (<70 mg/dL; <3.9 mmol/L) from BL | -1.6 [-138 to 131] | -47.7 [-71.9 to -17.6] | -84.4 [-101 to -50.3] | -19.9 [-174 to 135] | -58.9 [-65.9 to -27.9]
  Median Percent Change of Moderate Hypoglycemia Events (<60 mg/dL; <3.3 mmol/L) from BL | 14.6 [-314 to 498] | -65.3 [-84.5 to -18.8] | -94.8 [-106 to -58.0] | 20.8 [-499 to 540] | -64.4 [-74.1 to 7.30]
  Median Percent Change of Severe Hypoglycemia Events (<50 mg/dL; <2.8 mmol/L) from BL | -40.3 [-459 to 550] | -78.2 [-107 to 4.93] | -100 [-105 to -70.2] | -26.9 [-471 to 417] | -78.2 [-89.3 to -4.32]

6. Secondary Outcome: Median of Average Daily Percent Time With Overall, Moderate, and Severe Hypoglycemia by CGM at Baseline (BL) and End of Treatment (EOT)
Description: The median of average daily percent time in overall (<70 mg/dL [<3.9 mmol/L]), moderate (<60 mg/dL [3.3 mmol/L]), and severe (<50 mg/dL [2.8 mmol/L]) hypoglycemia at baseline (BL) and end of treatment (EOT) is reported.
Time Frame: 8 weeks
Population: Per Protocol Population
Measure: Median (95% Confidence Interval); unit: Daily Percent Time
Arm/Group | RZ358 Cohort 1 | RZ358 Cohort 2 | RZ358 Cohort 3 | RZ358 Cohort 4 | RZ358 Pooled
Number analyzed (Participants) | 4 | 8 | 7 | 3 | 22
Daily Percent Time
  Median Daily Percent Time in Overall Hypoglycemia (<70mg/dL; <3.9 mmol/L) at BL | 16.3 [7.83 to 24.8] | 20.3 [14.3 to 29.1] | 13.7 [-1.17 to 53.7] | 34.4 [-11.4 to 69.8] | 16.2 [15.2 to 31.2]
  Median Daily Percent Time in Overall Hypoglycemia (<70mg/dL; <3.9 mmol/L) at 8 Weeks (EOT) | 12.3 [1.28 to 19.6] | 6.68 [3.05 to 16.0] | 5.42 [-1.30 to 20.6] | 20.4 [-6.40 to 38.9] | 8.54 [6.73 to 14.6]
  Median Daily Percent Time in Moderate Hypoglycemia (<60 mg/dL; <3.3 mmol/L) at BL | 6.85 [1.53 to 11.5] | 8.75 [6.38 to 17.3] | 5.22 [-6.30 to 36.8] | 19.5 [-9.22 to 37.9] | 7.31 [6.19 to 18.4]
  Median Daily Percent Time in Moderate Hypoglycemia (<60 mg/dL; <3.3 mmol/L) at 8 Weeks (EOT) | 5.13 [0.05 to 9.39] | 3.25 [1.31 to 7.60] | 1.79 [-0.72 to 10.1] | 7.35 [-0.43 to 13.9] | 3.81 [3.06 to 6.73]
  Median Daily Percent Time in Severe Hypoglycemia (<50 mg/dL; < 2.8 mmol/L) at BL | 1.97 [-0.09 to 3.72] | 3.57 [2.12 to 8.17] | 1.12 [-3.70 to 13.9] | 3.03 [-4.08 to 11.2] | 2.56 [1.76 to 6.84]
  Median Daily Percent Time in Severe Hypoglycemia (<50 mg/dL; < 2.8 mmol/L) at 8 Weeks (EOT) | 1.27 [-0.216 to 3.04] | 1.05 [0.49 to 3.02] | 0.61 [-0.17 to 3.65] | 1.27 [-0.67 to 3.93] | 1.15 [1.01 to 2.33]

7. Secondary Outcome: Median Percent Change of Average Daily Percent Time With Overall, Moderate, and Severe Hypoglycemia by CGM From Baseline (BL)
Description: The average daily percent time in overall (<70 mg/dL [<3.9 mmol/L]), moderate (<60 mg/dL [3.3 mmol/L]), and severe (<50 mg/dL [2.8 mmol/L]) hypoglycemia is compared from baseline (BL) to end of treatment (EOT) and the median percent changes of those differences are reported.
Time Frame: 8 weeks
Population: Per Protocol Population
Measure: Median (95% Confidence Interval); unit: Percent Change
Arm/Group | RZ358 Cohort 1 | RZ358 Cohort 2 | RZ358 Cohort 3 | RZ358 Cohort 4 | RZ358 Pooled
Number analyzed (Participants) | 4 | 8 | 7 | 3 | 22
Percent Change
  Median Percent Change in Daily Percent Time in Overall Hypoglycemia (<70mg/dL; <3.9 mmol/L) from BL | -31.1 [-84.0 to 6.00] | -64.6 [-83.7 to -22.4] | -61.0 [-95.2 to -22.0] | -46.6 [-53.1 to -36.2] | -53.5 [-65.5 to -36.6]
  Median Percent Change in Daily Percent Time in Moderate Hypoglycemia (<60mg/dL; <3.3 mmol/L) from BL | -19.3 [-103 to 66.5] | -65.9 [-94.9 to -8.67] | -75.9 [-107 to 7.76] | -53.9 [-130 to 56.2] | -60.2 [-65.9 to -19.9]
  Median Percent Change in Daily Percent Time in Severe Hypoglycemia (<50 mg/dL; < 2.8 mmol/L) from BL | -21.9 [-299 to 447] | -74.4 [-120 to 54.0] | -85.0 [-164 to 178] | -60.7 [-213 to 173] | -64.8 [-66.6 to 68.8]

8. Secondary Outcome: Median of Average Daily Duration (Minutes) With Overall, Moderate, and Severe Hypoglycemia by CGM at Baseline (BL) and End of Treatment (EOT)
Description: The median of average duration (minutes) in overall (<70 mg/dL [<3.9 mmol/L]), moderate (<60 mg/dL [3.3 mmol/L] ), and severe (<50 mg/dL [2.8 mmol/L]) hypoglycemia by CGM at baseline (BL) and end of treatment (EOT) is reported.
Time Frame: 8 weeks
Population: Per Protocol Population
Measure: Median (95% Confidence Interval); unit: Daily Minutes in Hypoglycemia
Arm/Group | RZ358 Cohort 1 | RZ358 Cohort 2 | RZ358 Cohort 3 | RZ358 Cohort 4 | RZ358 Pooled
Number analyzed (Participants) | 4 | 8 | 7 | 3 | 22
Daily Minutes in Hypoglycemia
  Median Daily Duration (min) of Overall Hypoglycemia (<70 mg/dL; 3.9 mmol/L) at BL | 204 [107 to 301] | 266 [185 to 379] | 180 [8.77 to 675] | 472 [-177 to 966] | 214 [202 to 402]
  Median Daily Duration (min) of Overall Hypoglycemia (<70 mg/dL; 3.9 mmol/L) at 8 Weeks (EOT) | 158 [10.1 to 268] | 84.1 [36.5 to 208] | 76.7 [-19.5 to 293] | 287 [-93.6 to 554] | 99.1 [89.5 to 200]
  Median Daily Duration (min) of Moderate Hypoglycemia (<60 mg/dL; 3.3 mmol/L) at BL | 90.5 [21.8 to 141] | 113 [80.6 to 226] | 67.9 [-62.9 to 449] | 257 [-134 to 513] | 97.5 [83.7 to 232]
  Median Daily Duration (min) of Moderate Hypoglycemia (<60 mg/dL; 3.3 mmol/L) at 8 Weeks (EOT) | 65.8 [-4.32 to 130] | 35.7 [13.6 to 93.9] | 25.3 [-10.8 to 144] | 105 [-6.03 to 195] | 46.0 [39.3 to 90.6]
  Median Daily Duration (min) of Severe Hypoglycemia (<50 mg/dL; 2.8 mmol/L) at BL | 26.1 [-0.28 to 46.7] | 46.3 [26.1 to 105] | 14.3 [-37.5 to 159] | 39.3 [-61.1 to 152] | 32.7 [24.1 to 83.1]
  Median Daily Duration (min) of Severe Hypoglycemia (<50 mg/dL; 2.8 mmol/L) at 8 Weeks (EOT) | 15.00 [-5.07 to 41.2] | 14.8 [6.14 to 30.1] | 8.67 [-2.36 to 50.9] | 16.7 [-9.13 to 53.6] | 14.8 [12.2 to 29.0]

9. Secondary Outcome: Median Percent Change of Average Daily Duration (Minutes) With Overall, Moderate, and Severe Hypoglycemia by CGM From Baseline (BL)
Description: The average duration (minutes) in overall (<70 mg/dL [<3.9 mmol/L]), moderate (<60 mg/dL [3.3 mmol/L] ), and severe (<50 mg/dL [2.8 mmol/L]) hypoglycemia by CGM is compared from baseline (BL) to end of treatment (EOT) and the median percent changes of those differences are reported.
Time Frame: 8 weeks
Population: Per Protocol Population
Measure: Median (95% Confidence Interval); unit: Percent Change
Arm/Group | RZ358 Cohort 1 | RZ358 Cohort 2 | RZ358 Cohort 3 | RZ358 Cohort 4 | RZ358 Pooled
Number analyzed (Participants) | 4 | 8 | 7 | 3 | 22
Percent Change
  Median Percent Change in Daily Duration (min) of Overall Hypoglycemia (<70mg/dL; 3.9 mmol/L) from BL | -22.2 [-83.4 to 13.0] | -63.7 [-82.0 to -30.1] | -57.5 [-94.3 to -18.2] | -40.2 [-47.5 to -34.8] | -49.1 [-64.4 to -36.1]
  Median Percent Change in Daily Duration (min) of Moderate Hypoglycemia (<60mg/dL; 3.3mmol/L) from BL | 9.19 [-97.7 to 69.9] | -65.8 [-92.9 to -23.8] | -70.9 [-106 to 9.37] | -52.8 [-147 to 89.9] | -58.1 [-65.5 to -20.5]
  Median Percent Change in Daily Duration (min) of Severe Hypoglycemia (<50 mg/dL; 2.8 mmol/L) from BL | -18.6 [-272 to 400] | -77.0 [-107 to 7.36] | -81.2 [-160 to 171] | -59.8 [-325 to 357] | -63.0 [-66.2 to 61.3]

10. Secondary Outcome: Occurrence of Hypoglycemia During Fasting Challenge
Description: The occurrence of hypoglycemia during a 12 Hour fasting challenge.
Time Frame: 8 Weeks
Population: Per Protocol Population
Measure: Number; unit: participants
Arm/Group | RZ358 Cohort 1 | RZ358 Cohort 2 | RZ358 Cohort 3 | RZ358 Cohort 4 | RZ358 Pooled
Number analyzed (Participants) | 4 | 8 | 7 | 3 | 22
participants
  Number of patients able to complete fast at Baseline (n) | 3 | 2 | 0 | 0 | 5
  Number of patients able to complete fast at EOT (n) | 3 | 1 | 2 | 1 | 7

11. Secondary Outcome: Median of Average Hypoglycemia Events Per Day at Each of the Specified Glucose Thresholds by CGM at Baseline (BL) and End of Treatment (EOT)
Description: The median of average hypoglycemia events per day at each of the specified glucose thresholds [<70, <60, and <50 mg/dL (3.9, 3.3, and 2.8 mmol/L)], by CGM at baseline (BL) and end of treatment (EOT) is reported.
Time Frame: 8 weeks
Population: Per Protocol Population
Measure: Median (95% Confidence Interval); unit: Hypoglycemia Events Per Day
Arm/Group | RZ358 Cohort 1 | RZ358 Cohort 2 | RZ358 Cohort 3 | RZ358 Cohort 4 | RZ358 Pooled
Number analyzed (Participants) | 4 | 8 | 7 | 3 | 22
Hypoglycemia Events Per Day
  Median of Average Hypoglycemia Events Per Day <70mg/dL (3.9mmol/L) at BL | 3.00 [1.71 to 4.25] | 3.50 [2.40 to 4.30] | 2.46 [1.49 to 4.84] | 4.47 [2.18 to 6.22] | 3.37 [2.77 to 3.91]
  Median of Average Hypoglycemia Events Per Day <70mg/dL (3.9mmol/L) at 8 Weeks (EOT) | 2.37 [0.78 to 3.88] | 1.70 [0.93 to 3.78] | 2.33 [0.09 to 4.83] | 3.33 [-1.05 to 8.11] | 2.23 [1.72 to 3.37]
  Median of Average Hypoglycemia Events Per Day <60 mg/dL (3.3mmol/L) at BL | 1.73 [1.11 to 2.62] | 2.22 [1.59 to 3.52] | 1.77 [0.92 to 3.23] | 3.07 [0.30 to 5.53] | 2.00 [1.85 to 2.80]
  Median of Average Hypoglycemia Events Per Day <60 mg/dL (3.3mmol/L) at 8 Weeks (EOT) | 1.54 [0.60 to 2.53] | 1.06 [0.50 to 2.92] | 1.60 [-0.14 to 3.72] | 2.07 [-0.86 to 5.84] | 1.50 [1.15 to 2.48]
  Median Average Hypoglycemia Events Per Day <50mg/dL(2.8mmol/L) at BL | 0.91 [0.08 to 1.69] | 1.29 [0.61 to 2.33] | 0.79 [0.30 to 1.25] | 1.67 [-0.62 to 3.27] | 1.13 [0.77 to 1.47]
  Median Average Hypoglycemia Events Per Day <50mg/dL(2.8mmol/L) at 8 Weeks (EOT) | 0.74 [0.20 to 1.18] | 0.53 [0.23 to 1.40] | 0.60 [0.03 to 1.55] | 1.00 [-0.12 to 2.20] | 0.64 [0.54 to 1.09]

12. Secondary Outcome: Median Net Change of Average Hypoglycemia Events Per Day at Each of the Specified Glucose Thresholds by CGM From Baseline (BL)
Description: The average hypoglycemia events per day at each of the specified glucose thresholds [<70, <60, and <50 mg/dL (3.9, 3.3, and 2.8 mmol/L)], by CGM is compared from baseline (BL) to end of treatment (EOT) and the median net changes of those differences are reported.
Time Frame: 8 weeks
Population: Per Protocol Population
Measure: Median (95% Confidence Interval); unit: Events Per Day
Arm/Group | RZ358 Cohort 1 | RZ358 Cohort 2 | RZ358 Cohort 3 | RZ358 Cohort 4 | RZ358 Pooled
Number analyzed (Participants) | 4 | 8 | 7 | 3 | 22
Events Per Day
  Median Net Change of Average Hypoglycemia Events Per Day <70 mg/dL (3.9mmol/L) from BL | -0.47 [-1.98 to 0.69] | -1.41 [-2.04 to 0.04] | -1.49 [-3.76 to 2.34] | -1.14 [-3.48 to 2.14] | -1.05 [-1.67 to 0.08]
  Median Net Change of Average Hypoglycemia Events Per Day <60 mg/dL (3.3mmol/L) from BL | -0.32 [-1.48 to 0.89] | -0.82 [-1.57 to -0.13] | -0.63 [-2.48 to 1.90] | -0.39 [-1.82 to 0.97] | -0.61 [-1.14 to 0.12]
  Median Net Change of Average Hypoglycemia Events Per Day <50mg/dL(2.8mmol/L) from BL | -0.28 [-0.94 to 0.54] | -0.98 [-1.24 to -0.08] | -0.06 [-0.72 to 0.76] | -0.35 [-2.33 to 1.76] | -0.30 [-0.63 to 0.01]

13. Secondary Outcome: Median of Average 8-hour Overnight Percent Time in Glucose Target Range of 70-180mg/dL by CGM at Baseline (BL) and End of Treatment (EOT)
Description: The median of average 8-hour overnight (12am-8am) percent time within the glucose target range (70-180 mg/dL) at baseline (BL) and end of treatment (EOT) is reported.
Time Frame: 8 weeks
Population: Per Protocol Population
Measure: Median (95% Confidence Interval); unit: 8-hour Overnight Percent Time
Arm/Group | RZ358 Cohort 1 | RZ358 Cohort 2 | RZ358 Cohort 3 | RZ358 Cohort 4 | RZ358 Pooled
Number analyzed (Participants) | 4 | 8 | 7 | 3 | 22
8-hour Overnight Percent Time
  Median of Average 8h Overnight Percent Time in 70-180 mg/dL at BL | 80.8 [60.2 to 103] | 75.0 [70.1 to 86.6] | 82.1 [36.4 to 99.6] | 48.0 [-1.33 to 121] | 75.0 [63.1 to 83.1]
  Median of Average 8h Overnight Percent Time in 70-180 mg/dL at 8 Weeks (EOT) | 84.4 [68.2 to 103] | 81.1 [55.7 to 94.1] | 89.2 [62.5 to 96.0] | 73.8 [51.0 to 91.4] | 80.1 [69.9 to 85.6]

14. Secondary Outcome: Median Percent Change of Average 8-hour Overnight Percent Time in Glucose Target Range of 70-180mg/dL by CGM From Baseline (BL)
Description: The average 8-hour overnight (12am-8am) percent time within the glucose target range (70-180 mg/dL) is compared from baseline (BL) to end of treeatment (EOT) and the median percent change of that difference is reported.
Time Frame: 8 weeks
Population: Per Protocol Population
Measure: Median (95% Confidence Interval); unit: Percent Change
Arm/Group | RZ358 Cohort 1 | RZ358 Cohort 2 | RZ358 Cohort 3 | RZ358 Cohort 4 | RZ358 Pooled
Number analyzed (Participants) | 4 | 8 | 7 | 3 | 22
Percent Change | 7.59 [-4.71 to 15.8] | 3.67 [-28.6 to 22.4] | -2.64 [-59.1 to 211] | 44.1 [-58.7 to 116] | 4.22 [-11.1 to 66.9]

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Any untoward medical occurrence [i.e., any unfavorable and unintended sign (including abnormal lab findings), symptom or disease] which is either new or pre-existing but worsened in severity or frequency, whether or not it has a causal relationship to the study investigational (medicinal) products or procedures. Includes events w/ onset from the time of providing written informed consent until the EOS visit. AE may or may not be temporally or causally associated w/ the use of a study drug.
Arm/Group | RZ358 Cohort 1 | RZ358 Cohort 2 | RZ358 Cohort 3 | RZ358 Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8 | 0/8 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/8 | 1/8 | 0/3
Other Adverse Events (participants affected / at risk) | 2/4 | 7/8 | 5/8 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RZ358 Cohort 1 (N=4) | RZ358 Cohort 2 (N=8) | RZ358 Cohort 3 (N=8) | RZ358 Cohort 4 (N=3)
Hypoglycemia with LOC (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to the study drug. Patient had a medical history of hypoglycemia with LOC due to her background congenital HI.
Tonic-Clonic Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to study drug. Patient had a medical history of seizures.
Eosinophilic Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to study drug. Patient had medical history of pre-existing eosinophilia predominant leukocytosis.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RZ358 Cohort 1 (N=4) | RZ358 Cohort 2 (N=8) | RZ358 Cohort 3 (N=8) | RZ358 Cohort 4 (N=3)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion Site Reaction (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Medical Device Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalized tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychomotor Hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acanthosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sacral Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis Media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection, viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations include a small sample size (low statistical power), an open-label design (potential for bias due to lack of blinding), a short treatment period in a chronic disease, and a lack of ethnic diversity in study participants who have a rare pediatric disease. Additionally, the COVID-19 pandemic impacted the study by causing a delay in projected enrollment and study timelines. However, due to excess precaution taken, there was no impact on the overall execution/outcomes of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT04538989/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT04538989/SAP_001.pdf